CLINICAL TRIAL: NCT05469217
Title: The Effects of Fentanyl Abuse on Executive Function and Related Brain Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ariel University (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SMC-9459-22
Record Dates: First submitted 2022-07-20; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Fentanyl Dependence
Keywords: Fentanyl, gray matter, white matter, VBM, N-Back

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fentanyl dependent patients: 15 participants who were treated for fentanyl dependence in treatment centers in Israel
  Interventions: Other: fMRI brain imaging
- Control participants: Healthy control participants from the general public
  Interventions: Other: fMRI brain imaging

INTERVENTIONS:
Other: fMRI brain imaging — Structural MRI of gray and white matter, functional MRI during performance of the N-back task

SUMMARY:
There is a widespread abuse of prescription opioids and a dramatic increase in the availability of illicit opioids. These have created the "opioid epidemic" which is one of the most severe public health crisis in US History. Fentanyl, a synthetic opioid that is 50 to 100 times more potent than morphine, is a schedule II prescription drug used to treat severe pain. It is also a drug of abuse. Fentanyl is more likely to cause an overdose than is heroin because of its greater potency. In addition, it has a shorter half-life than most other opioids, causing the high to fade more quickly, requiring opioid drug abusers to inject more frequently, and increasing the risk of overdose. There is an increasing use of Fentanyl in Israel, and one of the treatment centers has reported that on average each month over the last year 10 patients that have used fentanyl were admitted. We propose to investigate executive function using established tasks such as the N-back and Go No Go tasks as well as structural brain imaging of gray matter volume and white matter tracts in 15 fentanyl abuse patients that will be compared with 15 healthy control participants.

DETAILED DESCRIPTION:
There is a widespread abuse of prescription opioids and a dramatic increase in the availability of illicit opioids. These have created the "opioid epidemic" which is one of the most severe public health crisis in US History (Skolnik, 2018; Volkow and Blanco, 2021). The magnitude of this epidemic is alarming. About 4% of the adult US population misuses prescription opioids, and in 2015, more than 33,000 deaths were attributable to overdose with licit and illicit opioids including Fentanyl (Skolnik, 2018). The number has increased in 2019 to 49,860 and in 2020 to over 93,000 deaths (Mattson et al., 2021; Lancet, 2021). The magnitude of the phenomenon is huge since there are over 125 million Americans suffering from either acute or chronic pain, and there is an urgent need for a long-term solution for controlling and ultimately eradicating this epidemic (Skolnik, 2018; France et al., 2021).

During the Covid-19 epidemic among individuals tested, there was an increase by 35% for non-prescribed fentanyl and 44% for heroin (Niles et al., (2021). Positive tests for non-prescribed fentanyl increased significantly among patients positive for other drugs: by 89% for specimens positive for amphetamines; 48% for benzodiazepines; 34% for cocaine; and 39% for opiates (Niles et al., 2021).

Fentanyl, a synthetic opioid that is 50 to 100 times more potent than morphine, is a schedule II prescription drug used to treat severe pain. It is also a drug of abuse. However, evidence from drug seizures by the US Drug Enforcement Agency indicates that fentanyl-related harm, overdose, and deaths in the United States are usually the result of illegally made fentanyl, sold through illicit drug markets for its euphoric effect. Fentanyl is more likely to cause an overdose than is heroin because of its greater potency. In addition, it has a shorter half-life than most other opioids, causing the high to fade more quickly, requiring opioid drug abusers to inject more frequently, and increasing the risk of overdose (Niles et al., 2021). The low production costs of fentanyl and its potency (50- fold compared to heroin) make it an attractive option to mix with heroin and illicit manufactured prescription opioids (Frank et al., 2017).

There is an increasing use of Fentanyl in Israel, and one of the treatment centers called "Haderech" in Ilabun has reported that on average each month over the last year 10 patients that have used fentanyl were admitted.

Currently, there are few studies that have investigated the effects of chronic long-term effects of opiate use on cognitive function and the brain. Steenbergen et al., (2019) have suggested that the mu-opioid system can influence higher-level cognitive function via modulation of evaluation, motivation, and control circuits dense in mu-opioid receptors, including the orbitofrontal cortex, basal ganglia, amygdala, anterior cingulate cortex, and the prefrontal cortex. They have proposed that opioids influence decision making and cognitive control by increasing the subjective value of reward and reducing aversive arousal (Steenbergn et al., 2019).

Initial research utilizing whole-brain neuroimaging techniques has identified structural differences in gray matter in opioid-dependent individuals although the results have been inconsistent. Wollman et al., (2017) have reported a meta-analysis of neuroimaging findings from 12 studies comparing opioid-dependent individuals to drug-naïve controls. Using Anisotropic Effect-Size Seed-Based d Mapping (AES-SDM) they have found that the fronto-temporal region, bilaterally, was the primary site of gray matter deficits associated with opioid use. Moderator analysis revealed that length of opioid use was negatively associated with gray matter in the left cerebellar vermis and the right Rolandic operculum, including the insula. Meta-regression revealed no remaining significant areas of gray matter reductions, except in the precuneus, following longer abstinence from opioids. They have concluded that Opioid-dependent individuals had significantly less gray matter in the frontal-cerebellar system that might be responsible for impulsivity, compulsive behaviors, and affective disturbances and the frontal-insular system that might account more for the cognitive and decision-making impairments.

To the best of our knowledge, there are no studies that have evaluated executive function impairment and gray matter and white matter structural changes as a result of fentanyl abuse. We propose to investigate executive function using established tasks such as the N-back task and structural brain imaging of gray matter volume and white matter tracts in 15 fentanyl abuse patients that will be compared with 15 healthy control participants. Patients will be recruited after treatment in the Israeli Ministry of Health treatment centers in Israel. The cognitive tasks and questionnaires evaluating drug abuse, anxiety and depression will be done by research assistants from the Dept. of Psychology and Behavioral science in Ariel University under responsibility of the co-principal investigator Prof. Aviv Weinstein. Structural fMRI imaging will be done in the dept. of diagnostic imaging in Tel Hashomer hospital under responsibility of the co-principal investigator Dr. Abigail Livny. We anticipate that this will be a pioneer study that may have major implications for our understanding of the long-term consequences of fentanyl abuse.

References France CP, Ahern GP, Averick S, Disney A, Enright HA, Esmaeli-Azad B, Federico A, Gerak LR, Husbands SM, Kolber B, Lau EY, Lao V, Maguire DR, Malfatti MA, Martinez G, Mayer BP, Pravetoni M, Sahibzada N, Skolnick P, Snyder EY, Tomycz N, Valdez CA, Zapf J. Countermeasures for Preventing and Treating Opioid Overdose. Clin Pharmacol Ther. 2021; 109(3):578-590. doi: 10.1002/cpt.2098. Epub 2020 Nov 29.

Frank RG, Pollack HA. Addressing the Fentanyl Threat to Public Health. The New England Journal of Medicine 2017; 376(7): 605-607.

The Lancet. A time of crisis for the opioid epidemic in the USA. Lancet. 2021; 24;398 (10297):277. doi: 10.1016/S0140-6736(21)01653-6.

Mattson CL, Tanz LJ, Quinn K, Kariisa M, Patel P, Davis NL. Trends and Geographic Patterns in Drug and Synthetic Opioid Overdose Deaths - United States, 2013-2019. MMWR Morb Mortal Wkly Rep 2021; 70:202-207. DOI: http://dx.doi.org/10.15585/mmwr.mm7006a4external icon Niles JK, Gudin J, Radcliff J, Kaufman HW. The Opioid Epidemic Within the COVID-19 Pandemic: Drug Testing in 2020. Popul Health Manag. 2021; 24(S1):S43-S51. doi: 10.1089/pop.2020.0230. Epub 2020 Oct 8.

Skolnick P. The Opioid Epidemic: Crisis and Solutions. Annu Rev Pharmacol Toxicol. 2018; 6;58:143-159. doi: 10.1146/annurev-pharmtox-010617-052534. Epub 2017 Oct 2.

van Steenbergen, H., Eikemo, M. & Leknes, S. The role of the opioid system in decision making and cognitive control: A review. Cogn Affect Behav Neurosci 19, 435-458 (2019). https://doi.org/10.3758/s13415-019-00710-6 Volkow ND, Blanco C. The changing opioid crisis: development, challenges and opportunities. Mol Psychiatry. 2021; 26(1):218-233. doi: 10.1038/s41380-020-0661-4. Epub 2020 Feb 4.

Wollman SC, Alhassoon OM, Hall MG, Stern MJ, Connors EJ, Kimmel CL, Allen KE, Stephan RA, Radua J. Gray matter abnormalities in opioid-dependent patients: A neuroimaging meta-analysis. Am J Drug Alcohol Abuse. 2017; 43(5):505-517. doi: 10.1080/00952990.2016.1245312. Epub 2016 Nov 3. PMID: 27808568.

ELIGIBILITY:
Inclusion Criteria: patients with Fentanyl dependence who have used the drug over the past year - Exclusion Criteria: Neurological impairment, Infectious diseases such as HIV/AIDS, pregnant women, underage, cocaine or alcohol abuse

Healthy control participants from the general public Exclusion Criteria: Neurological impairment, Infectious diseases such as HIV/AIDS, pregnant women, underage, cocaine or alcohol abuse

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 15 patients diagnosed with Fentanyl dependence will be recruited from treatment centers and 15 healthy control participants will be recruited from the general public
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gray matter volume in fMRI | 2 years
  Measures of gray matter volume in MRI
White matter volume in fMRI | 2 years
  Measures of white matter tracts in DTI in MRI
Executive function | 2 years
  Measures of brain activity on the N-Back task in fMRI

SECONDARY OUTCOMES:
N-back | 2 years
  Measures of performance on the N-Back task in fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Galia Zarfati, MD, Principal Investigator — Sheba Tel Hashomer Medical Center

IPD SHARING:
Plan to Share IPD: No